CLINICAL TRIAL: NCT05020691
Title: Non-invasive Ventilation in Covid-19 Respiratory Failure - Predicting Success: A Retrospective Observational Study to Determine Predictive Factors in the Success or Failure of Non-invasive Ventilation.
Brief Title: NIV in Covid-19 Respiratory Failure
Status: Terminated | Type: Observational
Why Stopped: Availability of research team limited by clinical workload (COVID-19)
Sponsor: National Heatlh Service Ayrshire and Arran (Other Government)
Responsible Party: Principal Investigator, Jamie Hooker, Senior Clinical Fellow, Intensive Care, National Heatlh Service Ayrshire and Arran
Other Study IDs: 298787
Record Dates: First submitted 2021-08-17; First posted 2021-08-25 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: COVID-19 Pneumonia
Keywords: Covid-19; HACOR; Non-Invasive Ventilation; CPAP
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective, single centre observational study to validate use of the HACOR score (Duan et al, 2017) in determining efficacy of non-invasive ventilation in Covid-19 respiratory failure.

DETAILED DESCRIPTION:
The investigators will retrospectively analyse medical records of patients with confirmed Covid-19 respiratory failure who received continuous positive airway pressure (CPAP) via facemask, as per clinician decision, in the High Dependency Unit (HDU) or Intensive Care Unit (ICU) of University Hospital Crosshouse between 1st March 2020 and 30th April 2021. By collecting baseline demographics and physiological data (including APACHE II and clinical frailty score) and calculating the HACOR score at initiation of CPAP, then at 1hr, 6hrs, 12hrs, 24hrs and 48hrs after initiating CPAP the investigators aim to validate use of the HACOR score in determining efficacy of NIV in Covid-19 respiratory failure. The investigators will also collect other variables (CRP and lymphocytes, lactate, mean arterial pressure, temperature) to determine if these factors have utility in predicting efficacy of NIV in Covid-19 respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed Covid-19 respiratory failure
2. NIV treatment instituted as per clinician decision
3. Admitted to HDU or ICU between 1/3/20 and 30/4/21

Exclusion Criteria:

1. Patients with immediate indication for invasive ventilation
2. Patients whose primary diagnosis was not Covid-19 respiratory failure, but received NIV in that time period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed Covid-19 respiratory failure treated with facemask CPAP in a district general hospital
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Escalation to Invasive Ventilation | Up to 6 months
  Number of patients who deteriorated after NIV commenced, requiring escalation to invasive ventilation
Death Due to Respiratory Failure | Up to 6 months
  Number of patients who deteriorated after NIV commenced, resulting in death due to respiratory failure
Clinical Improvement | Up to 6 months
  Number of patients who improved after NIV commenced, resulting in liberation from NIV (without requiring invasive ventilation)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Crosshouse, Kilmarnock, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duan J, Han X, Bai L, Zhou L, Huang S. Assessment of heart rate, acidosis, consciousness, oxygenation, and respiratory rate to predict noninvasive ventilation failure in hypoxemic patients. Intensive Care Med. 2017 Feb;43(2):192-199. doi: 10.1007/s00134-016-4601-3. Epub 2016 Nov 3. PMID 27812731